CLINICAL TRIAL: NCT02564549
Title: Multiparametric MRI-Based Active Surveillance to Avoid the Risks of Serial Biopsies in Men With Low-Risk Prostate Cancer (MAVERICK)
Brief Title: MRI-Based Active Surveillance to Avoid the Risks of Serial Biopsies in Men With Low-Risk Prostate Ca
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely and will not resume
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Massey Cancer Center (Other); Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MCC-14-10633; NCI-2015-01739 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 02147 (Other: Hunter Holmes McGuire VAMC)
Record Dates: First submitted 2015-09-28; First posted 2015-09-30 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma; Multiparametric MRI; Gleason's Score 6
Keywords: low risk prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (TRUS-guided biopsy) (Active Comparator): * Baseline and annual systematic TRUS-guided biopsy performed as per standard of care by urologists for a total of one baseline diagnostic biopsy and two active surveillance systematic biopsies.
  * mpMRI at the end of the 2nd year with targeted biopsy of any Prostate Imaging Reporting and Data System (PI-RADS) 4 or 5 lesion. Patients needing image- guided targeted biopsies will undergo this procedure by interventional radiology, which is a common standard of care at HHM VAMC.
  * Optional transperineal template biopsy of the prostate performed at end of 2nd year (month 25-30).
  * Patients will be followed, as per standard of care, for any potential infections from biopsies.
  * Annual PSA tests performed as per routine standard of care.
  Interventions: Procedure: TRUS-guided biopsy
- Group 2 (mpMRI with targeted biopsy) (Experimental): * Baseline systematic transrectal ultrasound-guided biopsy performed as per standard of care by urologists.
  * Baseline and annual mpMRI with targeted biopsy of any Prostate Imaging Reporting and Data System (PI-RADS) 4 or 5 lesion. Patients needing image- guided targeted biopsies will undergo this procedure by interventional radiology, which is a common standard of care at HHM VAMC.
  * Optional transperineal template biopsy of the prostate performed at end of 2nd year (month 25-30).
  * Patients will be followed, as per standard of care, for any potential infections from biopsies.
  * Annual PSA tests performed as per routine standard of care.
  Interventions: Procedure: mpMRI with targeted biopsy

INTERVENTIONS:
Procedure: TRUS-guided biopsy — Patients on the TRUS biopsy-based arm will undergo annual systematic biopsies without any MRI staging or guidance.
  Arms: Group 1 (TRUS-guided biopsy)
Procedure: mpMRI with targeted biopsy — Patients on the mpMRI- based arm will undergo annual mpMRI surveillance imaging, with image-guided targeted biopsies only as indicated by radiographic findings.
  Arms: Group 2 (mpMRI with targeted biopsy)

SUMMARY:
Phase II non-inferiority randomized trial of annual systematic biopsies versus mpMRI and targeted biopsies for men with low risk prostate cancer on active surveillance with any volume Gleason's Score 6, but no prior MRI imaging of the prostate.

DETAILED DESCRIPTION:
This is an unblinded, randomized trial of TRUS biopsy-based active surveillance versus mpMRI-based active surveillance. Patients on the TRUS biopsy-based arm will undergo annual systematic biopsies without any MRI staging or guidance. Patients on the mpMRI- based arm will undergo annual mpMRI surveillance imaging, with image-guided targeted biopsies only as indicated by radiographic findings.

ELIGIBILITY:
Inclusion Criteria:

* Prostate adenocarcinoma diagnosed by biopsy within 12 months prior to study registration.
* Gleason score ≤ 6
* PSA < 10 ng/mL
* Completed and documented history and physical addressing all inclusion/exclusion criteria.

Exclusion Criteria:

* A diagnosis of prostate adenocarcinoma on more than one set of prostate biopsies, on separate calendar dates.
* Previous MRI imaging of the prostate.
* Prior history of pelvic radiotherapy.
* Prior history of prostatectomy.
* Contraindication to prostate mpMRI (renal failure, hip prosthesis, pacemaker, etc).
* Contraindication to prostate biopsy via transrectal or transperineal approaches (including coagulopathy).
* Patients on testosterone replacement therapy who are unwilling to discontinue.
* Medical, psychological, or social condition that, in the opinion of the investigator, may increase the patient's risk or limit the patient's adherence with study requirements.
* Unable to understand, or unwilling to complete the informed consent process.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2016-06-28 (Actual); Study Completion 2017-10-13 (Actual)

PRIMARY OUTCOMES:
To asses the detection rate of Gleason score ≥ 4+3 in patients with low-risk prostate cancer who undergo transrectal ultrasound (TRUS) biopsy-based active surveillance (Group 1) versus patients who undergo mpMRI-based active surveillance (Group 2). | 3 years

SECONDARY OUTCOMES:
Percentage of patients in Group 1 versus Group 2 who remain on active surveillance from the time of randomization until the end of study participation. | 3 years
  To compare adherence with active surveillance requirements in Group 1 versus Group 2.
To compare the rate of biopsy-related infections in Group 1 versus Group 2. | 3 years
To compare the missed rate of occult Gleason score ≥ 4+3 by template biopsy at end of study in Group 1 versus Group 2. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Drew Moghanaki, MD, MPH, Principal Investigator — Massey Cancer Center
Locations (1):
- Hunter Holmes Mcguire Veteran Affairs Medical Center, Richmond, Virginia, United States